CLINICAL TRIAL: NCT03074708
Title: Zhujiang Hospital of the Southern Medical University
Brief Title: Application of 3D Visualization and 3D Printing in the Hepatobiliary and Pancreatic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Chihua Fang, Dr, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 001
Record Dates: First submitted 2016-01-29; First posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Liver Diseases; Pancreatic Diseases; Biliary Tract Diseases
Keywords: Three-Dimensional Image; Three Dimensional Printing
MeSH Terms: conditions — Liver Diseases; Pancreatic Diseases; Biliary Tract Diseases | interventions — Printing, Three-Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D visualization and 3D printing (Other): From January 2016 to December 2018,the clinical data of 200 patients with the hepatobiliary and pancreatic diseases will be collected.All the patients received abdominal CT scanning and 3D reconstruction. Then we used the 3D reconstruction model and the 3D printed model based on the 3D reconstruction model in the operation planning and the operation.The clinical data include operative time, intraoperative blood loss,and postoperative complications after surgery.
  Interventions: Other: 3D visualization and 3D printing

INTERVENTIONS:
Other: 3D visualization and 3D printing — From January 2016 to December 2018,the clinical data of 200 patients with the hepatobiliary and pancreatic diseases will be collected.All the patients received abdominal CT scanning and 3D reconstruction. Then we used the 3D reconstruction model and the 3D printed model based on the 3D reconstruction model in the operation planning and the operation.The clinical data include operative time, intraoperative blood loss,and postoperative complications after surgery.

SUMMARY:
Background:The aim of the study is to value the application of three-dimensional visualization and three-dimensional printing in the hepatobiliary and pancreatic surgery.Method：From January 2016 to December 2018,the clinical data of 200 patients with the hepatobiliary and pancreatic diseases will be collected.All the patients received abdominal CT scanning and 3D reconstruction. Then we used the 3D reconstruction model and the 3D printed model based on the 3D reconstruction model in the operation planning and the operation.The clinical data include operative time, intraoperative blood loss,and postoperative complications after surgery.

DETAILED DESCRIPTION:
From January 2016 to December 2018,the clinical data of 200 patients with the hepatobiliary and pancreatic diseases will be collected.All the patients received abdominal CT scanning and 3D reconstruction. Then we used the 3D reconstruction model and the 3D printed model based on the 3D reconstruction model in the operation planning and the operation.The clinical data include operative time, intraoperative blood loss,and postoperative complications after surgery.

ELIGIBILITY:
Inclusion Criteria:

* the hepatobiliary and pancreatic diseases

Exclusion Criteria:

* none of the hepatobiliary and pancreatic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
operative time | 1 year
  operative time

SECONDARY OUTCOMES:
intraoperative blood loss | 1 year
  intraoperative blood loss
postoperative complications after surgery | 1 year
  postoperative complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chihua Fang, MD, Study Chair — Zhujiang Hospital of The Southern Medical University
Locations (1):
- Zhujiang Hospital of The Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided